CLINICAL TRIAL: NCT05679921
Title: Pazopanib With or Without Pembrolizumab for Metastatic Soft Tissue Sarcoma: Open-label, Multicenter, Randomized, Phase 2 Trials
Brief Title: Pazopanib With or Without Pembrolizumab for Metastatic Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-1202
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Soft Tissue Sarcoma
Keywords: Sarcoma, Pembrolizumab, Pazopanib
MeSH Terms: conditions — Sarcoma | interventions — pembrolizumab; pazopanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PP1 (Experimental): pembrolizumab in combination with pazopanib
  Interventions: Drug: pembrolizumab, pazopanib
- PP2 (Experimental): pembrolizumab for patients progressing on pazopanib.
  Interventions: Drug: pembrolizumab, pazopanib

INTERVENTIONS:
Drug: pembrolizumab, pazopanib — Pembrolizumab will be given for a maximum of 2 years i.e. a total of 35 cycles of pembrolizumab with the q3 week dosing. Participants who complete study intervention after 2 years of pembrolizumab can be treated with pazopanib monotherapy based on physician's judgement. The duration of optional pembrolizumab crossover treatment will be maximum of 2 years i.e. a total of 35 cycles of pembrolizumab for patients progressing on pazopanib.

SUMMARY:
This is an open-label, randomized, phase II study to evaluate the clinical activity of pembrolizumab in combination with pazopanib compared to pazopanib monotherapy.

DETAILED DESCRIPTION:
Pembrolizumab will be given for a maximum of 2 years i.e. a total of 35 cycles of pembrolizumab with the q3 week dosing. Participants who complete study intervention after 2 years of pembrolizumab can be treated with pazopanib monotherapy based on physician's judgement. The duration of optional pembrolizumab crossover treatment will be maximum of 2 years i.e. a total of 35 cycles of pembrolizumab for patients progressing on pazopanib.

ELIGIBILITY:
Inclusion Criteria:

-

1. Histologically confirmed Soft Tissue Sarcoma(STS) progression to 1 or 2 (less than 3) prior chemotherapy : Exclude pazopanib-resistant subtype - embryonal rhabdomyosarcoma, chondrosarcoma, osteosarcoma, Ewing tumours, primitive neuroectodermal tumour, gastrointestinal stromal tumour, dermatofibrosarcoma protuberans, inflammatory myofibroblastic sarcoma, and liposarcoma
2. Age > 19 years, ≤80 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (within 7 days before screening)
4. Measurable disease by Response Evaluation Criteria in Solid Tumors Version 1.1
5. Adequate normal organ and marrow function as defined below -Hemoglobin ≥9.0 g/dL

   -Absolute neutrophil count (ANC) ≥ 1500 per mm3

   -Platelet count ≥ 100,000 per mm3

   -Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).

   -Aspartate Aminotransferase (AST, SGOT)/Alanine Aminotransferase (ALT, SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN

   -Creatinine≤1.5 x ULN

   -International normalized ratio (INR) OR prothrombin time (PT) and activated partial thromboplastin time (aPTT) : ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
6. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
7. A male or female participant must agree to use a contraception as detailed in Appendix 2 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
8. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 2 OR b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 2 during the treatment period and for at least 120 days after the last dose of study treatment.
9. Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

Exclusion Criteria:

1. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 14 days prior to the first dose of study drug
2. Any previous treatment with a Programmed Death-1(PD1) or Programmed Death-Ligand1(PD-L1) inhibitor, anti-PD-L2 agent, stimulatory/co-inhibitory T-cell receptor (eg. CTLA-4, OX-40, CD137), and/or pazopanib
3. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
4. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of Investigational Product(IP).

6. A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

7. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-Central Nervous System(CNS) disease.

8. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.

9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

10. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, urothelial cancer, or carcinoma in situ that have undergone potentially curative therapy are not excluded.

11. Has known active Central Nervous System (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable: without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention).

12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.

13. Has a history of or current(non-infectious) pneumonitis/interstitial lung disease that required steroids 14. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority. 15. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

* Note: Hepatitis B and C screening tests are not required unless:
* Known history of Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) infection
* As mandated by local health authority 16. Known active infection requiring systemic therapy.
* Active infection including tuberculosis
* Active hepatitis B (HBsAg reactive and HBV DNA is detected)
* Active hepatitis C (anti-HCV reactive and HCV RNA [qualitative] is detected)
* Human immunodeficiency virus infection 17. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

  18. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

  19. Has had an allogenic tissue/solid organ transplant. 20. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.

  21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

  22. Known or probable QT interval prolongation. 23. Any following history in past 6 months
* Coronary angioplasty or stent insertion, myocardial infarction, unstable angina, coronary artery bypass, New York Heart Association(NYHA) stage III or IV congestive heart failure, thromboembolism (stable patients on anticoagulation for at least 6 weeks can be enrolled), hemoptysis, brain hemorrhage or clinically significant gastrointestinal bleeding.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Rate (PFR) | 12 weeks
  Progression Free Rate (PFR)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 12 weeks
  Progression Free Survival (PFS)
Overall Response Rate (ORR) | 12 weeks
  Overall Response Rate (ORR)
Overall Survival(OS) | 4 months
  Overall Survival(OS)
Adverse Events(AE) | 6 months
  Adverse Events(AE)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No